CLINICAL TRIAL: NCT01571804
Title: Does Pregabalin Reduce the Sevoflurane Requirement During Laparoscopic Cholecystectomy? Mansoura University Hospitals Experience.
Brief Title: Pregabalin Reduce the Sevoflurane Requirement
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed R El Tahan, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R/49
Record Dates: First submitted 2012-03-31; First posted 2012-04-05 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Elective Laparoscopic Cholecystectomy; Sevoflurane Anesthesia
Keywords: Anesthesia; pregabalin; sevoflurane; laparoscopic cholecystectomy
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- pregabalin 150 mg group (Active Comparator): one capsule of pregabalin 150 mg and one placebo capsule
  Interventions: Drug: pregabalin
- pregabalin 300 mg group (Active Comparator): two capsules of pregabalin 150 mg
  Interventions: Drug: pregabalin
- placebo group (Placebo Comparator): to receive two identical placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — to receive two identical placebo capsules 1 hr before surgery
  Arms: placebo group
Drug: pregabalin — one capsule of pregabalin 150 mg and one placebo capsule 1 hr before surgery
  Arms: pregabalin 150 mg group
Drug: pregabalin — two capsules of pregabalin 150 mg 1 hr before surgery
  Arms: pregabalin 300 mg group

SUMMARY:
Preoperative administration of pregabalin would reduce the end tidal concentration of sevoflurane during laparoscopic cholecystectomy with added beneficial improving of the quality of postoperative analgesia.

DETAILED DESCRIPTION:
laparoscopic cholecystectomy is a painful and stressful surgical procedure. Pregabalin is a lipophilic structural analogue of the inhibitory γ-aminobutyric acid by binding to the presynaptic voltage-gated calcium channels that are widely distributed throughout the central and peripheral nervous system. Pregabalin has anticonvulsant, anxiolytic, sleep-modulating, anti-hyperalgesic, opioid-sparing6 and anti-allodynic properties through inhibition of the release of excitatory neurotransmitters such as glutamate, norepinephrine, serotonin, dopamine and substance P. These unique characteristics make pregabalin as a useful therapeutic for treating neuropathic pain and acute postoperative pain in several models of incisional injury and inflammatory conditions including laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists class I and II
* scheduled for elective laparoscopic cholecystectomy
* under sevoflurane anesthesia

Exclusion Criteria:

* communication barriers
* cardiovascular diseases
* renal diseases
* hepatic diseases
* endocrinal diseases
* neuropsychiatric diseases
* prolonged P-R interval
* pregnancy
* nursing
* hypersensitivity
* treated by pregabalin, antidepressant, anticonvulsants, opiates or benzodiazepines during the last week

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
changes in the end tidal sevoflurane concentrations | intraoperative every 15 min
  End-tidal concentrations of sevoflurane (Et-Sevo) were recorded every 15 min after intubation until the skin closure.

SECONDARY OUTCOMES:
hemodynamic parameters | before surgery, after the administration of the study capsules; intraoperative, an expected average of 2 hours, up to 24 after surgery
  heart rate and mean arterial blood pressure were recorded before (baseline), 45 min after the administration of the study capsules; every 15 min after intubation until the skin closure and every 15 min for the first hour after extubation.
intraoperative fentanyl supplementations | intraoperative, an expected average of 2 hours
  intraoperative fentanyl supplementations
quality of tracheal extubation | up to 24 after surgery
  The quality of tracheal extubation was evaluated using a 5 - points rating scale: 1, no coughing or straining; 2, very smooth, minimal coughing; 3, moderate coughing; 4, marked coughing or straining; and 5, poor extubation, very uncomfortable
postoperative cumulative morphine consumption | up to 24 after surgery
  postoperative cumulative morphine consumption
postoperative sedation and pain scores | up to 24 after surgery
  Postoperative pain VAS scores sedation (four-point verbal rating scores (VRS): awake, drowsy, rousable or deep sleep)
postoperative nausea and vomiting | up to 24 after surgery
  nausea and vomiting (0: no nausea; 1: nausea no vomiting; 2: nausea and vomiting)
awareness and recall | intraoperative, an expected average of 2 hours
  The patients were asked about intraoperative awareness and recall on the second postoperative day by asking three simple questions using standard interview "What was the last thing you remembered happening before you went to sleep? What is the first thing you remember happening on waking? Did you dream or have any other experiences whilst you were asleep?"

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospitals, Al Mansurah, DK, Egypt